CLINICAL TRIAL: NCT06068621
Title: Multicenter,Open Label,Phase 2 Clinical Study of Venetoclax Combined With CACAG Regimen in the Treatment of Newly Diagnosed Acute Myeloid Leukemia
Brief Title: Venetoclax Plus CACAG Regimen for Newly Diagnosed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: 940 Hospital of the People's Liberation Army Joint Logistic Support Force (Other); The General Hospital of Western Theater Command (Other); The General Hospital of Northern Theater Command (Other); The 960th Hospital of Joint Logistics Support Force of Chinese People's Liberation Army (Unknown); Air Force Military Medical University, China (Other); Yantai Yuhuangding Hospital (Other); People's Liberation Army (PLA) Strategic Support Force Characteristic Medical Center (Unknown); First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Daihong Liu, doctor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2023-056-01
Record Dates: First submitted 2023-09-29; First posted 2023-10-05 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; First Line Therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Venetoclax Combined With CACAG Regimen (Experimental): Venetoclax combined with CACAG regimen for newly diagnosed AML. Recipients were randomized and those entering the experimental group received azacytidine, cytarabine,aclacinomycin,chidamide,venetoclax and granulocyte colony-stimulating factor. Azacytidine was used as 75 mg/m2/day from day 1 to day 7. Cytarabine was used as 75-100 mg/m2 bid from day 1 to day 5. Aclacinomycin was used as 20 mg/day on days 1,3,5. Chidamide was used as 30 mg/day on days 1,4,8,11. Venetoclax was used as 400 mg/day from day 1 to day 14;Combined with posaconazole, reduced to 100 mg/day;Combined with voriconazole, reduced to 200 mg/day.Granulocyte colony-stimulating factor was used as 300 μg/day from day 0 until agranulocytosi recovery .
  Interventions: Drug: Azacytidine;Cytarabine;Aclacinomycin;Chidamide;Venetoclax;Granulocyte colony-stimulating factor
- "3+7" Regimen (Active Comparator): Idarubicin+cytarabine(IA) regimen or daunorubicin+cytarabine(DA) regimen for newly diagnosed AML.Recipients were randomized and those entering this group received IA or DA induction chemotherapy. With the IA regimen,recipients received idarubicin(8-10 mg/m2) for three days and cytarabine(75-100 mg/m2, every 12 hrs) for seven days. With the DA regimen,recipients received daunorubicin(60 mg/m2)for three days and cytarabine(75-100 mg/m2,every 12 hrs)for seven days.
  Interventions: Drug: "3+7"

INTERVENTIONS:
Drug: Azacytidine;Cytarabine;Aclacinomycin;Chidamide;Venetoclax;Granulocyte colony-stimulating factor — 1. Azacytidine (75 mg/m2/day, days 1 to 7).
  2. Cytarabine (75-100 mg/m2 bid, days 1 to 5).
  3. Aclacinomycin(20 mg/day, days 1,3,5).
  4. Chidamide (30 mg/day , days 1,4,8,11).
  5. Venetoclax (400 mg/day, days 1 to 14,Combined with posaconazole reduced to 100 mg/day,Combined with voriconazole reduced to 200 mg/day ).
  6. Granulocyte colony-stimulating factor (300 μg/day, day 0 until agranulocytosis recovery)
  Other Names: CACAG+VEN
  Arms: Venetoclax Combined With CACAG Regimen
Drug: "3+7" — IA regimen:
  1. Idarubicin (8-10 mg/m2) for 3 days .
  2. Cytarabine (75-100mg/m2, every 12 hrs) for 7 days.
  DA regimen:
  1. Daunorubicin(60 mg/m2) for 3 days.
  2. Cytarabine (75-100mg/m2, every 12 hrs) for 7 days.
  Other Names: IA or DA
  Arms: "3+7" Regimen

SUMMARY:
The purpose of this study is to compare the efficacy and safety of venetoclax combined with CACAG regimen with the traditional "3+7" regimen in the treatment of newly diagnosed acute myeloid leukemia.

DETAILED DESCRIPTION:
Despite the availability of hematopoietic stem cell transplantation and the emergence of many new therapeutic drugs, the prognosis of newly diagnosed acute myeloid leukemia is still poor.Over the past years, combination chemotherapy with anthracycline and standard dose cytarabine (standard "3+7" induction therapy) remains the standard induction. In order to improve the outcome of patients with de novo AML, we developed a venetoclax combined with CACAG regimen in the treatment of de novo AML. In this study, we intent to compare the efficacy and safety of venetoclax combined with CACAG regimen with the traditional "3+7" regimen in the treatment of newly diagnosed acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

Patients who are able to understand and willing to sign the informed consent form (ICF).

* All patients should aged 14 to75 years,no gender limitation.
* Patients who are newly diagnosed with AML(no M3).
* Liver function: ALT and AST≤2.5 times the upper limit of normal ,bilirubin≤2 times the upper limit of normal;
* Renal function: creatinine ≤the upper limit of normal;
* Patients without any uncontrolled infections , without organ dysfunction or without severe mental illness;
* The score of Eastern Cooperative Oncology Group (ECOG) is 0-2, and the predicted survival ≥ 4 months.
* Patients without severe allergic constitution.

Exclusion Criteria:

* Patients with allergy or contraindication to the study drug;
* Female patients who are pregnant or breast-feeding.
* Patients with a known history of alcohol or drug addiction on the basis that there could be a higher risk of non-compliance to study treatment;
* Patients with mental illness or other states unable to comply with the protocol;
* Less than 6 weeks after surgical operation of important organs.
* Liver function: ALT and AST>2.5 times the upper limit of normal ,bilirubin> 2 times the upper limit of normal;Renal function: creatinine >the upper limit of normal;
* The patient is not suitable for this clinical trial (poor compliance, substance abuse, etc.)

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) after 1 course of treatment | 1 months after the start of study treatment
  Defined as the percentage of participants achieving a best overall response of complete response (CR) or CR with incomplete blood count recovery (CRi).Biological characteristics exploratory studies were analyzed by single-cell sequencing and Atac-seq. Further, according to European LeukemiaNet risk group, we analyzed the outcomes of patients by molecular subtype as a sub-group analysis.

SECONDARY OUTCOMES:
Complete Remission (CR) Rate after 1 course of treatment | 2 months after study treatment
  Defined in accordance with the IWG Response Criteria in AML. Bone marrow blasts<5 percent; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count >1.0 x 109/L (1000/µL); platelet count >100 x 109/L (100,000/µL); independence of red cell transfusions.
Complete Remission (CR) Rate after 2 courses of treatment | after two courses of chemotherapy (each course is 28 days)
  Defined in accordance with the IWG Response Criteria in AML. Bone marrow blasts<5 percent; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count >1.0 x 109/L (1000/µL); platelet count >100 x 109/L (100,000/µL); independence of red cell transfusions.
Overall Response Rate (ORR) after 2 course of treatment | after two courses of chemotherapy (each course is 28 days)
  Defined as the percentage of participants achieving a best overall response of complete response (CR) or CR with incomplete blood count recovery (CRi).Biological characteristics exploratory studies were analyzed by single-cell sequencing and Atac-seq. Further, according to European LeukemiaNet risk group, we analyzed the outcomes of patients by molecular subtype as a sub-group analysis.
Rate of Minimal Residual Disease (MRD)-Negative Response | after two courses of chemotherapy (each course is 28 days)
  Percentage of participants who achieved MRD-negative response, defined as < 1 leukemia cell per 10,000 leukocytes as assessed by flow cytometry.
Event-free survival | 180 days after study treatment
  Defined as the time interval from treatment initiation to the occurrence of induction failure,relapse,or death,whichever came first.
Overall Survival (OS) | 180 days after study treatment
  Defined as the time from joining the clinical study to death due to any cause.
Treatment-related adverse events | From the first dose of study treatment to 30 days after the discontinuation of treatment
  Defined as adverse events that occurred from the first dose of study treatment to 30 days after the discontinuation of treatment.
Early death | Within 30 days of the start of the first course of treatment
  Defined as death within 30 days of chemotherapy.
Disease-free survival | 180 days after study treatment
  Defined as the time interval from disease remission to the occurrence of relapse or death,whichever came first.

CONTACTS AND LOCATIONS:
Overall Officials: Daihong Liu, doctor, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China